CLINICAL TRIAL: NCT05976087
Title: Improving Grasp Function in People With Sensorimotor Impairments by Combining Electrical Stimulation With a Robotic Hand Orthosis
Acronym: SENSIBLE-EXO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrea Cimolato (Other)
Responsible Party: Sponsor-Investigator, Andrea Cimolato, Study coordinator, ETH Zurich
Organization: ETH Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-010428
Record Dates: First submitted 2023-07-19; First posted 2023-08-04 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Spinal Cord Injuries; Traumatic Brain Injury
Keywords: sensorimotor; TENS; FES; exoskeleton; wearable robotics
MeSH Terms: conditions — Stroke; Spinal Cord Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Device: SensoExo

INTERVENTIONS:
Device: SensoExo — combination of sensory feedback and the use of soft exoskeleton

SUMMARY:
Hand motor and sensory impairments resulting from neurological disorders or injuries affect more than 50 million individuals worldwide. Conditions such as stroke, spinal cord injury (SCI), and traumatic brain injury (TBI) can cause long-term hand impairments, greatly impacting daily activities and social integration. Since traditional physiotherapy has limited effectiveness in rehabilitation, assistive devices helping in performing in daily activities have emerged as a necessary solution. Soft exoskeletons offer advantages as they are more comfortable and adaptable for the user, but they often struggle to generate sufficient force. On the other hand, electrical stimulation garments, like e-sleeves, show promise by stimulating nerves and muscles in the forearm. However, achieving precise and stable movement control remains challenging due to difficulties in electrode placement for targeted stimulation. Furthermore, none of the currently available devices are capable of artificially restoring lost sensation in users' hands, limiting their ability to manipulate with fragile objects.

Recognizing these limitations, our study proposes a solution that combines a standard hand soft exoskeleton with: (i) electrical stimulation to the fingers' flexor and extensor muscles to generate artificial muscle contractions synchronized with the exoskeleton motion, compensating for the lack of gripping force, and (ii) electrical stimulation to the nerves to artificially restore the lost sensation of touch, enabling users to receive feedback on the force they are applying when interacting with the environment. The investigators refer to this proposed combination as Sensible-Exo.

To achieve this goal, our project aims to evaluate the functional improvements in assistive and rehabilitative scenarios using SensoExo in comparison to use only the exoskeleton or having no support at all. The exoskeleton will be coupled with an electrical stimulating sleeve capable of delivering non-invasive electrical stimulation in the form of Functional Electrical Stimulation (FES) and Transcutaneous Electrical Nerve Stimulation (TENS). A glove with embedded force and bending sensors will be used to modulate the electrical stimulation. Additionally, apart from studying the enhancement of functional tasks, the investigators will explore improvements in body perception, representation, and multi-sensory integration. Indeed, the investigators also aim at identifying the way patients perceive their body by means of ad-hoc virtual reality assessments that has been developed. Before each assessment patient will perform some predefined movement in virtual reality to familiarize with it and increase embodiment.

During the study, participants will perform a range of tasks based on their residual abilities, including motor tasks (e.g., grab and release, Toronto Rehabilitation Institute Hand Function Test, grip force regulation test, virtual egg test), cognitive tasks (dual tasks), and assessments of body representation and perception. Some of these tasks will be conducted in Virtual Reality environments, both with and without active stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Impairment of the motor and sensory functions of the hand in chronic stage
* The subject should have good proximal arm function (i.e. good shoulder abduction and elevation)

Exclusion Criteria:

* Cognitive and communication deficits impairment
* Prior or current psychological diseases such as borderline, schizophrenia, Depression or Maniac Depression
* Major comprehension and memory deficits
* Pregnancy
* Epilepsy
* Pacemaker
* Cybersickness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Range of Motion with electrical stimulation and without no electrical stimulation | up to one month before; thorugh study completition (average 1 month); up to one month after
  Range of motion will be measured and compared among conditions
Change in the area with tactile feedback in the hand with electrical stimulation and with no electrical stimulation | up to one month before; thorugh study completition (average 1 month); up to one month after
  Semmes-Weinstein Monofilament Test will be used to assess the residual tactile feedback
Change in functional tasks performance with sensory feedback and without sensory feedback quantified by the number of successful grasp and release tasks | up to one month before; thorugh study completition (average 1 month); up to one month after
  Number of successful transportation of objects over an obstacle
Change between functional tasks with sensory feedback and with no sensory feedback in number of virtual egg successful grasping | up to one month before; thorugh study completition (average 1 month); up to one month after
  Number of successful transportations of fragile objects over an obstacle
Change between functional tasks with sensory feedback and with no sensory feedback in grasping force | up to one month before; thorugh study completition (average 1 month); up to one month after
  Grasping forces will be assessed during functional performance of the subjects
Change between tasks with sensory feedback and with no sensory feedback in arm joints kinemtics | up to one month before; thorugh study completition (average 1 month); up to one month after
  Joint kinematics measurements will be measured with motion capture systems during functional performance of the subjects

SECONDARY OUTCOMES:
Change in experienced physical, mental, and social effects | up one week before first session and up one week after last session
  Neuro-QuL measurement system will be as assessment tool
Change in Proprioceptive drift between different conditions | up one week before first session and up one week after last session
  To measure embodiment subjects will be asked after VR sessions to indicate where they feel their arm without looking at the limb in real world. This is a measure of embodiment.
Change in Telescoping measures between different conditions | up one week before first session and up one week after last session
  To measure embodiment subjects will be asked after VR sessions to indicate how long they feel their arm without looking at the limb in real world. This is a measure of embodiment.
Change from baseline performance between tasks accomplished with sensory feedback and with no sensory feedback in Embodiment | up one week before first session and up one week after last session
  Embodiment will be measured with questionnaires (from -3 to +3, +3 totally agrees; two questions are from 1 to 10 (to measure vividness, where 10 is max vividness) and from 1 to 100 (to measure prevalence, where 100 is max duration of the embodiment feeling))
Measures of self-body representation | up one week before first session; thorugh study completition (average 1 month); up one week after last session
  This will be measured in virtual reality by means of ad-hoc Body Landmark test. This is a body representation measurements.
Measures of body-space representation | up one week before first session; thorugh study completition (average 1 month); up one week after last session
  This will be measured in virtual reality by means of ad-hoc Hand Peri personal Space test. This is a body representation measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Stanisa Raspopovic, PhD, Principal Investigator — ETH Zurich
Locations (1):
- Neuroengineering Lab, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dannenbaum RM, Dykes RW. Sensory loss in the hand after sensory stroke: therapeutic rationale. Arch Phys Med Rehabil. 1988 Oct;69(10):833-9. PMID 3178450
- [Background] Carey LM, Matyas TA, Oke LE. Sensory loss in stroke patients: effective training of tactile and proprioceptive discrimination. Arch Phys Med Rehabil. 1993 Jun;74(6):602-11. doi: 10.1016/0003-9993(93)90158-7. PMID 8503750
- [Background] Finnerup NB, Johannesen IL, Fuglsang-Frederiksen A, Bach FW, Jensen TS. Sensory function in spinal cord injury patients with and without central pain. Brain. 2003 Jan;126(Pt 1):57-70. doi: 10.1093/brain/awg007. PMID 12477697
- [Background] Fujimoto ST, Longhi L, Saatman KE, Conte V, Stocchetti N, McIntosh TK. Motor and cognitive function evaluation following experimental traumatic brain injury. Neurosci Biobehav Rev. 2004 Jul;28(4):365-78. doi: 10.1016/j.neubiorev.2004.06.002. PMID 15341032
- [Background] Dannenbaum RM, Jones LA. The assessment and treatment of patients who have sensory loss following cortical lesions. J Hand Ther. 1993 Apr-Jun;6(2):130-8. doi: 10.1016/s0894-1130(12)80294-8. PMID 8343879
- [Background] Kwakkel G, Kollen BJ, van der Grond J, Prevo AJ. Probability of regaining dexterity in the flaccid upper limb: impact of severity of paresis and time since onset in acute stroke. Stroke. 2003 Sep;34(9):2181-6. doi: 10.1161/01.STR.0000087172.16305.CD. Epub 2003 Aug 7. PMID 12907818
- [Background] Wade DT. Measuring arm impairment and disability after stroke. Int Disabil Stud. 1989 Apr-Jun;11(2):89-92. doi: 10.3109/03790798909166398. PMID 2698395
- [Background] Fuhrer MJ, Rintala DH, Hart KA, Clearman R, Young ME. Relationship of life satisfaction to impairment, disability, and handicap among persons with spinal cord injury living in the community. Arch Phys Med Rehabil. 1992 Jun;73(6):552-7. PMID 1622304
- [Background] Noreau L, Fougeyrollas P. Long-term consequences of spinal cord injury on social participation: the occurrence of handicap situations. Disabil Rehabil. 2000 Mar 10;22(4):170-80. doi: 10.1080/096382800296863. PMID 10798305
- [Background] Butzer T, Lambercy O, Arata J, Gassert R. Fully Wearable Actuated Soft Exoskeleton for Grasping Assistance in Everyday Activities. Soft Robot. 2021 Apr;8(2):128-143. doi: 10.1089/soro.2019.0135. Epub 2020 Jun 18. PMID 32552422
- [Background] Beekhuizen KS. New perspectives on improving upper extremity function after spinal cord injury. J Neurol Phys Ther. 2005 Sep;29(3):157-62. doi: 10.1097/01.npt.0000282248.15911.38. PMID 16398948
- [Background] Lambercy O, Dovat L, Yun H, Wee SK, Kuah CW, Chua KS, Gassert R, Milner TE, Teo CL, Burdet E. Effects of a robot-assisted training of grasp and pronation/supination in chronic stroke: a pilot study. J Neuroeng Rehabil. 2011 Nov 16;8:63. doi: 10.1186/1743-0003-8-63. PMID 22087842
- [Background] Marquez-Chin C, Popovic MR. Functional electrical stimulation therapy for restoration of motor function after spinal cord injury and stroke: a review. Biomed Eng Online. 2020 May 24;19(1):34. doi: 10.1186/s12938-020-00773-4. PMID 32448143
- [Background] Ciancibello J, King K, Meghrazi MA, Padmanaban S, Levy T, Ramdeo R, Straka M, Bouton C. Closed-loop neuromuscular electrical stimulation using feedforward-feedback control and textile electrodes to regulate grasp force in quadriplegia. Bioelectron Med. 2019 Nov 1;5:19. doi: 10.1186/s42234-019-0034-y. eCollection 2019. PMID 32232108
- [Background] Prochazka A, Gauthier M, Wieler M, Kenwell Z. The bionic glove: an electrical stimulator garment that provides controlled grasp and hand opening in quadriplegia. Arch Phys Med Rehabil. 1997 Jun;78(6):608-14. doi: 10.1016/s0003-9993(97)90426-3. PMID 9196468